CLINICAL TRIAL: NCT04429451
Title: Phase I/II Clinical Trial of 4SCAR-PSMA T Cell Therapy Targeting PSMA Positive Malignancies
Brief Title: PSMA-specific CAR-T Cell Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Shenzhen Children's Hospital (Other Government); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20003
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: PSMA Positive Tumors or Tumor Tissues
Keywords: chimeric antigen receptor; adoptive T cell transfer; PSMA; Prostate cancer; Tumor microenvironment; CAR
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR-PSMA Cell Therapy for PSMA positive tumor (Experimental): Infusion of 4SCAR-PSMA T cells at 10^6 cells/kg body weight via IV
  Interventions: Biological: 4SCAR-PSMA T cells

INTERVENTIONS:
Biological: 4SCAR-PSMA T cells — Infusion of 4SCAR-PSMA T cells at 10^6 cells/kg body weight via IV

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of PSMA-specific CAR-T cell therapy in patients with PSMA positive tumor. Another goal of the study is to learn more about the function of the PSMA CAR-T cells and their persistency in the patients.

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA) is expressed in normal prostate and is upregulated in prostate tumor. Therefore, PSMA is a promising target for antigen-specific immunotherapy in patients with prostate cancer. However, it has been reported that PSMA expression is not restricted to prostate cancer and PSMA is often enriched in the tumor stromal environment. By immunostaining, we found that PSMA is expressed in a variety of solid tumors, including brain tumor, neuroblastoma and some lymphoma tumor tissues.

This study aims to use T cells obtained directly from the patient, which can be genetically modified to express PSMA-specific chimeric antigen receptor (CAR). The CAR molecules enable the T cells to recognize and kill tumor cells or tumor stromal tissues through the recognition of a surface antigen, PSMA. This study will evaluate the side effects and the best dose of anti-PSMA CAR-T cells to target PSMA positive tumors and tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with tumors have received standard first-line therapy and have been judged to be non-respectable, metastatic, progressive or recurrent.
2. The expression status of PSMA antigens in the tumor tissue will be determined for eligibility. Positive expression is defined by PMSA antibody staining results based on immunohistochemistry or flow cytometry analyses.
3. Body weight greater than or equal to 10 kg.
4. Age: ≥1 year and ≤ 75 years of age at the time of enrollment.
5. Life expectancy: at least 8 weeks.
6. Prior Therapy:

   There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less.
7. Participant must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection.
8. At least 7 days must have elapsed since the completion of therapy with a biologic agent, targeted agent, tyrosine kinase inhibitor or a metronomic non-myelosuppressive regimen.
9. At least 4 weeks must have elapsed since prior therapy that included a monoclonal antibody.
10. At least 1 week since any radiation therapy at the time of study entry.
11. Karnofsky/jansky score of 60% or greater.
12. Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent.
13. Pulse Ox greater than or equal to 90% on room air.
14. Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
15. Renal function: Patients must have serum creatinine less than 3 times upper limit of normal.
16. Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
17. Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease does not have hematologic toxicity.
18. For all patients enrolled in this study, themselves or their parents or legal guardians must sign an informed consent and assent.

Exclusion Criteria:

1. Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, or greater than grade 2 hematologic toxicity.
2. Untreatable central nervous system (CNS) metastasis: Patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
3. Previous treatment with other genetically engineered PSMA-specific CAR T cells or antibody therapy.
4. Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
5. Patients who require systemic corticosteroid or other immunosuppressive therapy.
6. Evidence of tumor potentially causing airway obstruction.
7. Inability to comply with protocol requirements.
8. Insufficient CAR T cells availability.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 3 year
  Determine the toxicity profile the 4SCAR-PSMA cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 1 year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
The expansion and persistence of 4SCAR-PSMA T cells | 1 year
  Scale of CAR copies and tumor burden (for efficacy)
Survival time of the patients | 3 year
  The survival time of the patients treated with the 4SCAR-PSMA T cells, including progression free survival (PFS) and overall survival (OS) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - The Seventh Affilliated Hospital of Sun Yat-Sen University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No